CLINICAL TRIAL: NCT02848313
Title: An Open-Label, Phase 1 Clinical Study to Evaluate the Safety and Tolerability of Subcutaneous Elamipretide in Subjects With Intermediate Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPIAM-101
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Intervention Model Description: Both arms received 40 mg dose of elamipretide administered once daily as a 1.0mL SC injection.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermediate AMD - HRD without GA (Experimental): Participants had one 1 eye with intermediate age-related macular degeneration with high-risk drusen without geographic atrophy [GA]), i.e. the presence of either at least 1 large (≥125 μm) druse or multiple medium-size (63-124 μm) drusen.
  Participants received 40 mg dose of elamipretide administered once daily as a 1.0mL SC injection.
  Interventions: Drug: Elamipretide
- Intermediate AMD with NCGA (Experimental): Participants had 1 eye with intermediate AMD with noncentral geographic atrophy [NCGA]; i.e. evidence of GA with cumulative area ≥1.27 mm2 (approximately 0.5 disc area[DA]) by fundus autofluorescence (FAF) that spared the fovea (defined as retinal pigment epithelium (RPE) and outer retina intact by spectral-domain optical coherence tomography [SD-OCT]).
  Participants in this arm also received 40 mg dose of elamipretide administered once daily as a 1.0mL SC injection.
  Interventions: Drug: Elamipretide

INTERVENTIONS:
Drug: Elamipretide — 40 mg dose of elamipretide administered once daily as a 1.0mL SC injection.
  Other Names: MTP-131; Bendavia

SUMMARY:
This is an open-label, Phase 1 single-center study in approximately 40 subjects who have 1 eye with intermediate AMD, including a high-risk drusen without geographic atrophy (GA) subgroup and a noncentral GA subgroup. Eligible subjects will receive 40 mg of elamipretide administered as a once daily 1.0 mL subcutaneous injection for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

For this study, only 1 eye of an eligible subject will be included and designated as the study eye. However, all specified ophthalmic testing will be performed on both eyes at each time point. A potential subject must meet the following criteria to be eligible for inclusion in the study:

Intermediate AMD - noncentral GA disease group:

1. Adults ≥ 55 years of age with 1 eye with intermediate AMD - noncentral GA.
2. No evidence of choroidal neovascularization (active or prior history) in the study eye.
3. Geographic atrophy may be multifocal, but the cumulative GA lesion size must be:

   1. ≥ 1.27 mm2 (approximately ≥ 0.5 DA) and ≤ 10.16 mm2 (approximately ≤ 4 DA).
   2. Must reside completely within the FAF imaging field (field 2 to 30-degree image centered on the fovea).
4. Presence of measurable hyperautofluorescence adjacent to the discrete foci of GA.

   OR

   Intermediate AMD - high-risk drusen without GA disease group:
5. ≥ 55 years of age with one eye with intermediate AMD - high-risk drusen without GA.
6. High-risk drusen is defined as presence of either at least 1 large (≥ 125 µm) druse or multiple medium-size (between 63 and 124 µm) drusen.

   General (both disease groups):
7. Able to provide informed consent and willing to comply with all study visits and examinations.
8. Women of childbearing potential who are not pregnant or nursing and have a negative serum pregnancy test at screening.
9. Best-corrected visual acuity assessed by ETDRS letters ≥ 55 letters (Snellen equivalent ≥ 20/70).
10. Low-luminance visual acuity deficit (defined as difference between BCVA and LL visual acuity) > 5 letters.
11. Has at least two Low-Luminance Questionnaire sub scale results, in which one of the abnormal subscales is either general dim light vision or dim light reading.
12. The fellow eye may have intermediate AMD without noncentral GA (i.e., high-risk drusen), intermediate AMD with noncentral GA, NV AMD, or central GA. Ongoing treatment with antiangiogenic therapies in the fellow eye is allowable.
13. No evidence of visually significant cataract OR pseudophakia without evidence of posterior capsular opacity.
14. Sufficiently clear ocular media, adequate pupillary dilation, fixation to permit quality fundus imaging, and able to cooperate sufficiently for adequate ophthalmic visual function testing and anatomic assessment.
15. Able to administer SC study drug solution as demonstrated at screening or able to have a care provider or appropriate designee who can administer the study drug (i.e., a capable family member or home health nursing aide).
16. If of childbearing potential or in a relationship with a partner of childbearing potential, are able to abstain from sex or use acceptable contraception during the study and for 3 months after dosing.

    1. For men: Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the subject. The subject also agrees to use an acceptable method of contraception should they become sexually active. Subjects must use a condom with spermicide from the date of informed consent until at least 3 months after the last dose of study drug. Periodic abstinence (e.g.calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
    2. For women: abstinence is only acceptable when it is in line with the preferred and usual lifestyle of the subject. The subject agrees to use an acceptable method of contraception should they become sexually active. Maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy (the vasectomy procedure must have been conducted at least 60 days before the Screening visit or confirmed via sperm analysis), barrier method (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream AND either hormonal contraception (oral, implanted, or injectable) or an intrauterine device or system are acceptable methods.
17. Ability and willingness to undertake all scheduled visits and assessments.

Exclusion Criteria:

A subject with study eye who meets any of the following criteria will be excluded from the study:

Ocular conditions - study eye

1. Age-related macular degeneration with any evidence of central GA (i.e., involving the fovea).
2. Atrophic retinal disease because of causes other than AMD.
3. Presence or diagnosis of exudative AMD or choroidal neovascularization in the study eye.
4. History of diabetic retinopathy (a history of diabetes mellitus without retinopathy is not a criterion for exclusion).
5. Presence of vitreous hemorrhage.
6. History of retinal detachment or macular hole (stage 3 or 4) in the study eye.
7. Presence of macular pucker.
8. History of uncontrolled glaucoma, defined as advanced cup-to-disc ratio > 0.7 and IOP > 25, with or without topical antihypertensive eye drops; treatment of ocular hypertension or controlled glaucoma are not criteria for exclusion.
9. History of advanced guttae indicative of Fuchs endothelial dystrophy.
10. Presence of visually significant cataract OR presence of significant posterior capsular opacity in the setting of Pseudophakia.
11. Presence of significant keratopathy that would cause scattering of light or alter visual function, especially in LL conditions.
12. Ocular incisional surgery (including cataract surgery) in the study eye within 3 months (i.e. 90 days) before Day 1.
13. Aphakia.
14. History of vitrectomy surgery, submacular surgery, or any vitreoretinal surgery.
15. Prior treatment with Visudyne ® (verteporfin), external-beam radiation therapy (for intraocular conditions), or transpupillary thermotherapy.
16. History of prophylactic subthreshold laser treatment for retinal disease.
17. Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection, anti-angiogenic drugs, or device implantation) in the study eye.

    Ocular conditions - either eye
18. Active uveitis and/or vitritis (grade trace or above) in either eye.
19. History of idiopathic or autoimmune-associated uveitis in either eye.
20. Active, infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.

    Systemic conditions
21. Known to be immunocompromised or receiving systemic immunosuppression.
22. Any disease or medical condition that in the opinion of the Investigator would prevent the subject from participating in the study or might confound study results.
23. Estimated glomerular filtration rate < 30 mL/minute, by MDRD.
24. Presence or history of clinically significant allergy disease requiring treatment, as judged by the Investigator. Hay fever is allowed unless it is active.

    General
25. Participation in other investigational drug or device clinical trials within 30 days before enrollment, or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion.
26. History of allergy to fluorescein that is not amenable to treatment.
27. Inability to comply with study or follow-up procedures.
28. Inability to obtain color fundus photograph, FAF, and fluorescein angiography of sufficient quality to be analyzed and interpreted.
29. History of allergic reaction to the investigational drug or any of its components.
30. Current use of or likely need for any excluded medication.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Cousins, MD, Principal Investigator — Duke University School of Medicine / Dept. of Ophthalmology (Duke Eye Center)
Locations (1):
- Duke University School of Medicine / Dept. of Ophthalmology (Duke Eye Center), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Risk Drusen (HRD): The HRD cohort was defined as the presence of either at least 1 large (≥125 μm) druse or multiple medium-size (63-124 μm) drusen in one eye. Subjects had to have 1 eye with intermediate AMD (high-risk drusen [HRD] without geographic atrophy [GA]).
- NCGA (Noncentral GA): The NCGA cohort was defined as evidence of GA with cumulative area ≥1.27 mm2 (approximately 0.5 disc area) by fundus autofluorescence (FAF) that spared the fovea (defined as retinal pigment epithelium and outer retina intact by spectral-domain optical coherence tomography [SD-OCT]). Subjects had to have 1 eye with intermediate AMD with noncentral GA [NCGA]
Period: Overall Study
Arm/Group | High-Risk Drusen (HRD) | NCGA (Noncentral GA)
Started | 21 | 19
Completed | 18 | 15
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to follow up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Risk Drusen (HRD) | NCGA (Noncentral GA) | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (8.54) | 76.0 (8.22) | 73.3 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking Status [Count of Participants; unit: Participants]
  Never smoker | 13 | 8 | 21
  Former smoker | 8 | 11 | 19
  Current smoker | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Standard Luminance Best-corrected Visual Acuity (BCVA)
Description: Change from Baseline in Mean Standard Luminance Best-corrected Visual Acuity (BCVA) at 4 meters, letters from Baseline to Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 28.
Time Frame: Day 0 (Baseline to Day 7, and to Weeks 4, 8, 12, 16, 20, 24, and 28.
Population: All participants for whom Standard Luminance BCVA was measured.
Measure: Mean (Standard Deviation); unit: letters
Groups:
- AMD-High-Risk Drusen (HRD): The HRD cohort was defined as the presence of either at least 1 large (≥125 μm) druse or multiple medium-size (63-124 μm) drusen in one eye. Subjects had to have 1 eye with intermediate AMD (high-risk drusen [HRD] without geographic atrophy [GA]).
- AMD-NCGA (Noncentral GA): The NCGA cohort was defined as evidence of GA with cumulative area ≥1.27 mm2 (approximately 0.5 disc area) by fundus autofluorescence (FAF) that spared the fovea (defined as retinal pigment epithelium and outer retina intact by spectral-domain optical coherence tomography [SD-OCT]). Subjects had to have 1 eye with intermediate AMD with noncentral GA [NCGA]
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 19
letters
  Day 7 | 0.810 (4.8746) | 0.526 (4.1281)
  Week 4: number analyzed (Participants) | 21 | 18
  Week 4 | 2.762 (5.5759) | 1.833 (5.0904)
  Week 8: number analyzed (Participants) | 20 | 18
  Week 8 | 1.950 (4.4066) | 1.556 (6.2987)
  Week 12: number analyzed (Participants) | 20 | 16
  Week 12 | 1.150 (5.5845) | 1.438 (5.4156)
  Week 16: number analyzed (Participants) | 19 | 16
  Week 16 | 2.789 (5.8933) | 2.813 (5.5883)
  Week 20: number analyzed (Participants) | 19 | 16
  Week 20 | 3.842 (4.1401) | 1.438 (5.7847)
  Week 24: number analyzed (Participants) | 19 | 15
  Week 24 | 3.579 (6.3972) | 4.600 (5.0681)
  Week 28: number analyzed (Participants) | 18 | 15
  Week 28 | 1.333 (10.4881) | 3.667 (5.8023)

2. Secondary Outcome: Change From Baseline in Mean Low Luminance Best-Corrected Visual Acuity (LLBCVA)
Description: Change from Baseline in Mean Low Luminance Best-Corrected Visual Acuity (LLBCVA) from Baseline (Day 0) to Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 28.
Time Frame: Baseline to Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 28.
Population: All participants for whom Standard Luminance BCVA was measured.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 19
letters
  Day 7 | 2.714 (5.3399) | 1.105 (8.4518)
  Week 4: number analyzed (Participants) | 21 | 18
  Week 4 | 2.762 (4.8673) | 5.000 (5.5413)
  Week 8: number analyzed (Participants) | 20 | 18
  Week 8 | 2.800 (6.2205) | 4.167 (4.2183)
  Week 12: number analyzed (Participants) | 20 | 16
  Week 12 | 2.150 (6.6986) | 4.688 (4.5858)
  Week 16: number analyzed (Participants) | 19 | 16
  Week 16 | 5.158 (7.3126) | 4.875 (5.9203)
  Week 20: number analyzed (Participants) | 19 | 16
  Week 20 | 5.632 (7.4923) | 5.438 (5.8875)
  Week 24: number analyzed (Participants) | 19 | 15
  Week 24 | 5.632 (7.7832) | 5.400 (7.8540)
  Week 28: number analyzed (Participants) | 18 | 15
  Week 28 | 2.556 (14.2095) | 3.733 (8.1545)

3. Secondary Outcome: Change From Baseline in Mean Dark Adaptometry
Description: Change from Baseline in Mean Dark Adaptometry from Baseline to Week 24- at 0% 25%, 50%, 75% Bleach Level. Dark adaptometry, used to evaluate night blindness by measuring the absolute thresholds of rod sensitivity, was performed within 14 days before Day 0 and at all in-person visits except for Day 7. Dark adaptation is the delayed recovery of light sensitivity in darkness following prior light exposure (photobleaching). The observed and change from baseline recovery scores (in minutes) for each bleach level (0%, 25%, 50%, and 75%) were summarized descriptively for each eye at each visit and were presented in a listing. Shorter recovery times are better than longer recovery times.
Time Frame: Baseline (Day 0) and Week 24
Population: All participants for whom Dark Adaptometry was measured at Baseline and Week 24 at 0% 25%, 50%, 75% Bleach Level.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 19
minutes
  0% Bleach Level | -11.553 (10.3229) | 3.543 (5.0140)
  25% Bleach Level: number analyzed (Participants) | 12 | 8
  25% Bleach Level | 0.409 (4.2798) | 8.3302 (0.000)
  50% Bleach Level: number analyzed (Participants) | 8 | 6
  50% Bleach Level | 0.000 (0.0000) | -3.263 (7.9935)
  75% Bleach Level: number analyzed (Participants) | 12 | 6
  75% Bleach Level | 1.562 (5.3936) | -3.048 (9.1675)

4. Secondary Outcome: Mean Treatment Compliance (%) of Administration of Subcutaneous Elamipretide
Description: Mean percentage of treatment compliance of administration of subcutaneous elamipretide. The number of injections (diary) and vials used was used to compute % compliance over the duration of the subject's participation in the trial. Percentage can range from 0-100%, where 0% means the participant followed the correct dosing 0% of the time, and 100% compliance means the participant followed the correct dosing 100% of the time, with a higher % meaning a better outcome.
Time Frame: Baseline through Week 28
Population: All participants for whom compliance was measured.
Measure: Mean (Standard Deviation); unit: % of compliance in study dosing
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 19
% of compliance in study dosing | 98.4 (4.04) | 97.3 (6.70)

5. Secondary Outcome: Mean Number of Home Health Visits to Administer Elamipretide
Description: Mean Number of Home Health Visits Necessary for Participant or Caregiver to Learn How to Administer Elamipretide
Time Frame: Baseline (Day 0) through Week 24
Population: All participants and caregivers whom administered elamipretide injections.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 19
visits | 2.2 (0.54) | 2.5 (1.02)

6. Secondary Outcome: Change From Baseline in Mean Area of Geographic Atrophy by Fundus Autofluorescence
Description: Change from Baseline in Mean Area of Geographic Atrophy (GA) by Fundus Autofluorescence (FAF) at Week 24. Fluorescein angiography (FA) was used to examine the circulation of the retina and choroid using fluorescein dye and a specialized camera to trace the dye. Fundus autofluorescence imaging of the retinal pigment epithelium and neurosensory retina was performed within 14 days of Day 0 and at every visit with the exception of Day 0 and Day 7. Atrophy is characterized by loss of the retinal pigment epithelium (RPE), overlying photoreceptors and underlying choriocapillaris. Greater area affected means a worse outcome than smaller area affected.
Time Frame: Baseline (Day 0) to Week 24
Population: All participants for whom Geographic Atrophy by Fundus Autofluorescence was measured at Week 24.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 0 | 12
mm^2
  Week 12: number analyzed (Participants) | 0 | 11
  Week 12 |  | 0.264 (0.1641)
  Week 24 |  | 0.503 (0.4914)

7. Secondary Outcome: Change From Baseline in Mean Area of Geographic Atrophy as Measured by Spectral-Domain Optical Coherence Tomography (SD-OCT)
Description: Change from Baseline in Mean Area of Geographic Atrophy by Sector as measured by Spectral-Domain Optical Coherence Tomography (SD-OCT) at Week 24
Time Frame: Baseline to Week 24
Population: All participants for whom geographic atrophy by SD-OCT was measured.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 0 | 15
mm^2
  Center Sector |  | 0.02 (0.048)
  Inner Superior |  | 0.05 (0.096)
  Inner Nasal |  | 0.04 (0.059)
  Inner Inferior |  | 0.02 (0.073)
  Inner Temporal |  | 0.05 (0.097)
  Outer Superior |  | 0.08 (0.116)
  Outer Nasal |  | 0.06 (0.114)
  Outer Inferior |  | 0.05 (0.146)
  Outer Temporal |  | 0.08 (0.129)
  Total ETDRS grid |  | 0.45 (0.607)

8. Secondary Outcome: Change From Baseline in Mean Reading Acuity Test: With Standard Luminance
Description: Change from Baseline in Mean Reading Acuity Test: Mean Critical Print Size with Standard Luminance in Weeks 4, 8, 12, 16, 20, 24 and 28 as measured by the Logarithm of the Minimum Angle of Resolution LogMAR chart. Scores range from -0.3 to 1.0, where higher number means worse acuity/worse outcome, a lower number means better acuity/better outcome.
Time Frame: Baseline and Weeks 4, 8, 12, 16 20, 24 and 28
Population: All participants for whom Mean Critical Print Size (logMAR) with Standard Luminance was measured
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 18
units on a scale
  Week 4 | -0.04 (0.121) | -0.03 (0.091)
  Week 8: number analyzed (Participants) | 20 | 18
  Week 8 | -0.08 (0.111) | -0.02 (0.115)
  Week 12: number analyzed (Participants) | 20 | 16
  Week 12 | -0.10 (0.156) | -0.02 (0.098)
  Week 16: number analyzed (Participants) | 19 | 16
  Week 16 | -0.11 (0.151) | -0.06 (0.115)
  Week 20: number analyzed (Participants) | 19 | 16
  Week 20 | -0.12 (0.126) | -0.01 (0.109)
  Week 24: number analyzed (Participants) | 19 | 15
  Week 24 | -0.11 (0.152) | -0.02 (0.126)
  Week 28: number analyzed (Participants) | 18 | 15
  Week 28 | -0.04 (0.201) | 0.01 (0.173)

9. Secondary Outcome: Change From Baseline in Mean Reading Acuity Test: Low Luminance
Description: Change from Baseline in Mean Reading Acuity Test: Mean Critical Print Size with Low Luminance in Weeks 4, 8, 12, 16, 20, 24 and 28 as measured by the Logarithm of the Minimum Angle of Resolution LogMAR chart. Scores range from -0.3 to 1.0, where higher number means worse acuity/worse outcome, a lower number means better acuity/better outcome.
Time Frame: Assessed at screening, baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 28
Population: All participants for whom Mean Critical Print Size (logMAR) with Low Luminance was measured at baseline and Week 4 through Week 28.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 11
units on a scale
  Week 4: number analyzed (Participants) | 21 | 10
  Week 4 | -0.11 (0.170) | -0.09 (0.088)
  Week 8: number analyzed (Participants) | 20 | 11
  Week 8 | -0.16 (0.179) | -0.10 (0.253)
  Week 12: number analyzed (Participants) | 20 | 10
  Week 12 | -0.21 (0.177) | -0.20 (0.236)
  Week 16: number analyzed (Participants) | 19 | 10
  Week 16 | -0.25 (0.209) | -0.16 (0.232)
  Week 20: number analyzed (Participants) | 19 | 10
  Week 20 | -0.29 (0.184) | -0.14 (0.171)
  Week 24: number analyzed (Participants) | 19 | 9
  Week 24 | -0.28 (0.174) | -0.11 (0.209)
  Week 28: number analyzed (Participants) | 18 | 9
  Week 28 | -0.24 (0.238) | -0.10 (0.194)

10. Secondary Outcome: Change From Baseline in National Eye Institute Visual Function Questionnaire-39 (VFQ-39) Score Standard Luminance
Description: Change from baseline (Day 0) at Week 12, 24 and 28. National Eye Institute Visual Function Questionnaire-39 (VFQ-39) score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at baseline (Day 0), Week 12, Week 24 and Week 28
Population: All participants for whom the VFQ-39 was measured at Week 12 and Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 20 | 16
score on a scale
  Week 12 Color Vision | 8.8 (18.63) | 10.9 (20.35)
  Week 12 Composite | 7.6 (7.47) | 5.5 (8.90)
  Week 12 Dependency | 1.9 (10.94) | 2.0 (14.02)
  Week 12 Distance Activities | 7.0 (8.13) | 4.6 (12.19)
  Week 12 Driving: number analyzed (Participants) | 20 | 13
  Week 12 Driving | 10.0 (12.85) | 0.6 (13.38)
  Week 12 General Health | 1.4 (8.98) | 1.9 (9.33)
  Week 12 General Vision | 5.3 (11.18) | 7.2 (14.02)
  Week 12 Mental Health | 9.3 (13.79) | 9.1 (14.63)
  Week 12 Near Activities | 8.2 (10.43) | 2.4 (11.51)
  Week 12 Ocular Pain | 7.5 (20.84) | 3.1 (9.68)
  Week 12 Peripheral Vision | 12.5 (19.02) | 7.8 (19.83)
  Week 12 Role Difficulties | 5.9 (12.25) | 5.9 (26.37)
  Week 12 Social Functioning | 7.5 (8.51) | 5.2 (18.48)
  Week 24 Color Vision: number analyzed (Participants) | 19 | 15
  Week 24 Color Vision | 11.8 (22.62) | 11.7 (26.50)
  Week 24 Composite: number analyzed (Participants) | 19 | 15
  Week 24 Composite | 9.2 (9.19) | 7.0 (9.38)
  Week 24 Dependency: number analyzed (Participants) | 19 | 15
  Week 24 Dependency | 2.3 (14.61) | 6.7 (10.94)
  Week 24 Distance Activities: number analyzed (Participants) | 19 | 15
  Week 24 Distance Activities | 8.4 (11.11) | 4.7 (16.13)
  Week 24 Driving: number analyzed (Participants) | 19 | 13
  Week 24 Driving | 14.5 (14.66) | 0.6 (10.46)
  Week 24 General Health: number analyzed (Participants) | 19 | 15
  Week 24 General Health | -0.3 (9.01) | 3.3 (10.21)
  Week 24 General Vision: number analyzed (Participants) | 19 | 15
  Week 24 General Vision | 8.7 (12.78) | 6.3 (13.69)
  Week 24 Mental Health: number analyzed (Participants) | 19 | 15
  Week 24 Mental Health | 9.5 (17.55) | 7.7 (9.80)
  Week 24 Near Activities: number analyzed (Participants) | 19 | 15
  Week 24 Near Activities | 9.8 (11.00) | 5.6 (13.84)
  Week 24 Ocular Pain: number analyzed (Participants) | 19 | 15
  Week 24 Ocular Pain | 5.9 (19.26) | 5.0 (14.02)
  Week 24 Peripheral Vision: number analyzed (Participants) | 19 | 15
  Week 24 Peripheral Vision | 17.1 (16.78) | 15.0 (18.42)
  Week 24 Role Difficulties: number analyzed (Participants) | 19 | 15
  Week 24 Role Difficulties | 6.9 (11.58) | 5.8 (17.27)
  Week 24 Social Functioning: number analyzed (Participants) | 19 | 15
  Week 24 Social Functioning | 6.6 (10.96) | 5.6 (15.64)
  Week 28 Color Vision: number analyzed (Participants) | 18 | 15
  Week 28 Color Vision | 12.5 (17.68) | 5.0 (28.66)
  Week 28 Composite: number analyzed (Participants) | 18 | 15
  Week 28 Composite | 7.9 (14.04) | 4.3 (10.46)
  Week 28 Dependency: number analyzed (Participants) | 18 | 15
  Week 28 Dependency | 1.7 (17.91) | -1.3 (20.07)
  Week 28 Distance Activities: number analyzed (Participants) | 18 | 15
  Week 28 Distance Activities | 5.7 (16.92) | 7.1 (13.95)
  Week 28 Driving: number analyzed (Participants) | 17 | 11
  Week 28 Driving | 12.3 (12.54) | 0.8 (9.47)
  Week 28 General Health: number analyzed (Participants) | 18 | 15
  Week 28 General Health | 4.2 (10.18) | 4.0 (9.20)
  Week 28 General Vision: number analyzed (Participants) | 18 | 15
  Week 28 General Vision | 8.6 (16.25) | 3.7 (12.60)
  Week 28 Mental Health: number analyzed (Participants) | 18 | 15
  Week 28 Mental Health | 9.4 (19.84) | 5.7 (10.50)
  Week 28 Near Activities: number analyzed (Participants) | 18 | 15
  Week 28 Near Activities | 6.0 (20.17) | 1.7 (12.63)
  Week 28 Ocular Pain: number analyzed (Participants) | 18 | 15
  Week 28 Ocular Pain | 7.6 (20.17) | 0.0 (14.94)
  Week 28 Peripheral Vision: number analyzed (Participants) | 18 | 15
  Week 28 Peripheral Vision | 15.3 (21.25) | 13.3 (20.85)
  Week 28 Role Difficulties: number analyzed (Participants) | 18 | 15
  Week 28 Role Difficulties | 4.2 (21.00) | 5.4 (20.03)
  Week 28 Social Functioning: number analyzed (Participants) | 18 | 15
  Week 28 Social Functioning | 5.6 (17.85) | 3.3 (10.82)

11. Secondary Outcome: Change From Baseline in Mean Low Luminance Questionnaire (LLQ) Score
Description: Change from baseline (Day 0) at Week 12, Week 24, and Week 28 in LLQ score. The LLQ is a 32-item questionnaire with six subscales related to low luminance settings: driving, mobility, extreme lighting, general dim lighting, and peripheral vision. Each question is scored on a scale ranging from 0, or maximal difficulty, to 100, or no difficulty in low luminance settings. Higher scores mean better functioning. The questions are assigned to different subscales and are averaged to generate one score per subscale. After weighting each subscale for the number of questions, the weighted subscales are averaged to generate a composite LLQ score.
Time Frame: Baseline (Day 0), Week 12, and Week 24 and Week 28
Population: All participants for whom Low-Luminance visual function by the Visual Function Questionnaire was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 21 | 16
score on a scale
  Week 12 Control questions: number analyzed (Participants) | 20 | 16
  Week 12 Control questions | 10.5 (15.47) | -2.3 (9.86)
  Week 12 Dim light reading: number analyzed (Participants) | 20 | 16
  Week 12 Dim light reading | 9.7 (12.58) | 4.3 (13.05)
  Week 12 Driving or riding in car: number analyzed (Participants) | 20 | 16
  Week 12 Driving or riding in car | 12.2 (16.41) | 3.9 (10.92)
  Week 12 General dim light vision: number analyzed (Participants) | 20 | 16
  Week 12 General dim light vision | 11.9 (13.26) | 6.9 (12.62)
  Week 12 Light transitions and glare: number analyzed (Participants) | 20 | 16
  Week 12 Light transitions and glare | 9.3 (15.07) | 6.3 (13.35)
  Week 12 Mobility: number analyzed (Participants) | 20 | 16
  Week 12 Mobility | 6.7 (11.66) | 6.3 (10.32)
  Week 12 Other Activities of Daily Living (ADLs): number analyzed (Participants) | 20 | 16
  Week 12 Other Activities of Daily Living (ADLs) | 11.5 (18.36) | 10.2 (15.29)
  Week 12 Peripheral vision: number analyzed (Participants) | 20 | 16
  Week 12 Peripheral vision | 16.3 (19.49) | 3.9 (17.51)
  Week 24 Control questions: number analyzed (Participants) | 21 | 15
  Week 24 Control questions | 7.2 (12.56) | 0.7 (12.47)
  Week 24 Dim light reading: number analyzed (Participants) | 19 | 15
  Week 24 Dim light reading | 15.8 (14.34) | 7.1 (11.30)
  Week 24 Driving or riding in car: number analyzed (Participants) | 19 | 15
  Week 24 Driving or riding in car | 16.4 (18.77) | 4.2 (14.11)
  Week 24 General dim light vision: number analyzed (Participants) | 19 | 15
  Week 24 General dim light vision | 15.6 (15.17) | 7.7 (12.10)
  Week 24 Light transitions and glare: number analyzed (Participants) | 19 | 15
  Week 24 Light transitions and glare | 17.4 (13.98) | 6.7 (13.71)
  Week 24 Mobility: number analyzed (Participants) | 19 | 15
  Week 24 Mobility | 9.6 (20.27) | 2.8 (16.57)
  Week 24 Other Activities of Daily Living (ADLs): number analyzed (Participants) | 19 | 15
  Week 24 Other Activities of Daily Living (ADLs) | 17.8 (17.95) | 10.4 (20.82)
  Week 24 Peripheral vision: number analyzed (Participants) | 19 | 15
  Week 24 Peripheral vision | 17.8 (20.12) | 5.8 (24.03)
  Week 28 Control Questions: number analyzed (Participants) | 21 | 15
  Week 28 Control Questions | 3.2 (18.44) | 0.2 (14.25)
  Week 28 Dim light reading: number analyzed (Participants) | 21 | 15
  Week 28 Dim light reading | 12.2 (19.70) | 7.1 (12.47)
  Week 28 Driving or riding in car: number analyzed (Participants) | 21 | 15
  Week 28 Driving or riding in car | 10.8 (23.85) | 4.3 (14.34)
  Week 28 General dim light vision: number analyzed (Participants) | 21 | 15
  Week 28 General dim light vision | 11.7 (19.43) | 3.3 (10.73)
  Week 28 Light transitions and glare: number analyzed (Participants) | 21 | 15
  Week 28 Light transitions and glare | 15.0 (14.75) | 5.3 (14.07)
  Week 28 Mobility: number analyzed (Participants) | 21 | 15
  Week 28 Mobility | 7.4 (23.02) | -1.1 (14.39)
  Week 28 Other Activities of Daily Living: number analyzed (Participants) | 21 | 15
  Week 28 Other Activities of Daily Living | 12.2 (23.82) | 3.8 (13.73)
  Week 28 Peripheral Vision: number analyzed (Participants) | 21 | 15
  Week 28 Peripheral Vision | 13.9 (20.06) | 5.0 (15.53)

12. Secondary Outcome: Change From Baseline in Mean Mesopic Light Sensitivity
Description: Change from baseline in mean mesopic light sensitivity for Weeks, 4, 8, 12, 16, 20, and 24 as assessed by microperimetry for number of loci <25dB and <14dB. Mesopic microperimetry, used to measure retinal sensitivity, was performed within 14 days before Day 0 and at all in-person visits except for Day 7.
Time Frame: Baseline (Day 0) and Weeks 4,8,12,16,20,and 24
Population: All participants for whom mean mesopic light sensitivity was measured.
Measure: Mean (Standard Deviation); unit: loci
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 20 | 17
loci
  Number of loci <25dB Week 4: number analyzed (Participants) | 20 | 14
  Number of loci <25dB Week 4 | 0.6 (6.08) | 0.6 (1.79)
  Number of loci <25dB Week 8: number analyzed (Participants) | 18 | 15
  Number of loci <25dB Week 8 | 1.3 (8.21) | 0.7 (1.94)
  Number of loci <25dB Week 12: number analyzed (Participants) | 17 | 17
  Number of loci <25dB Week 12 | 0.5 (7.87) | 0.1 (3.09)
  Number of loci <25dB Week 16: number analyzed (Participants) | 16 | 14
  Number of loci <25dB Week 16 | 0.9 (8.56) | 0.1 (2.35)
  Number of loci <25dB Week 20: number analyzed (Participants) | 17 | 15
  Number of loci <25dB Week 20 | -1.2 (5.88) | -0.1 (1.44)
  Number of loci <25dB Week 24: number analyzed (Participants) | 17 | 13
  Number of loci <25dB Week 24 | -0.5 (8.27) | -0.1 (3.45)
  Number of loci <14dB Week 4: number analyzed (Participants) | 4 | 13
  Number of loci <14dB Week 4 | 0.3 (0.3) | 1.7 (1.7)
  Number of loci <14dB Week 8: number analyzed (Participants) | 5 | 14
  Number of loci <14dB Week 8 | -1.4 (3.65) | 1.7 (4.89)
  Number of loci <14dB Week 12: number analyzed (Participants) | 4 | 16
  Number of loci <14dB Week 12 | 1.3 (10.05) | 3.2 (5.90)
  Number of loci <14dB Week 16: number analyzed (Participants) | 4 | 13
  Number of loci <14dB Week 16 | -2.5 (2.38) | 1.5 (5.01)
  Number of loci <14dB Week 20: number analyzed (Participants) | 5 | 14
  Number of loci <14dB Week 20 | -0.2 (6.14) | 1.5 (4.88)
  Number of loci <14dB Week 24: number analyzed (Participants) | 4 | 12
  Number of loci <14dB Week 24 | -0.3 (8.30) | 3.3 (5.82)

13. Secondary Outcome: Change From Baseline in Mean Retinal Pigment Epithelium - Drusen Complex (RPEDC) Thickness as Measured by SD-OCT
Description: Change from baseline in mean retinal pigment epithelium - drusen complex (RPEDC) thickness as Measured by SD-OCT by sector at Week 24
Time Frame: Baseline (Day 0) and Week 24
Population: All participants for whom RPEDC) thickness as Measured by SD-OCT by sector at Baseline and Week 24
Measure: Mean (Standard Deviation); unit: um
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 19 | 15
um
  Center | 0.57 (5.147) | 0.38 (4.137)
  Inner Superior | 1.29 (3.699) | -0.85 (2.389)
  Inner Nasal: number analyzed (Participants) | 19 | 5
  Inner Nasal | 1.43 (3.143) | -0.83 (2.801)
  Inner Inferior | 0.72 (4.393) | -0.82 (3.798)
  Inner temporal | 1.00 (3.680) | -0.34 (2.897)
  Outer Superior | 0.34 (2.279) | -0.10 (1.580)
  Outer Nasal | 0.34 (2.301) | -0.09 (1.919)
  Outer Inferior | -0.19 (2.356) | -0.04 (2.023)
  Outer Temporal | 0.25 (2.672) | -0.04 (1.594)
  Total ETDRS | 0.39 (1.885) | -0.25 (1.590)

14. Secondary Outcome: Change From Baseline in Mean Retinal Pigment Epithelium-Drusen Complex Volume
Description: Change from baseline in mean Retinal Pigment Epithelium-Drusen Complex volume at Week 24 by sector
Time Frame: Baseline (Day 0) to Week 24
Population: All participants for whom the retinal pigment epithelium-drusen complex volume was measured
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | AMD-High-Risk Drusen (HRD) | AMD-NCGA (Noncentral GA)
Number analyzed (Participants) | 19 | 15
mm^3
  Center | 0.00 (0.004) | 0.00 (0.003)
  Inner superior | 0.00 (0.006) | -0.00 (0.004)
  Inner nasal | 0.00 (0.005) | -0.00 (0.004)
  Inner inferior | 0.00 (0.007) | -0.00 (0.006)
  Inner temporal | 0.00 (0.006) | -0.00 (0.005)
  Outer superior | 0.00 (0.012) | -0.00 (0.008)
  Outer nasal | 0.00 (0.012) | -0.00 (0.010)
  Outer inferior | -0.00 (0.012) | -0.00 (0.011)
  Outer temporal | 0.00 (0.014) | -0.00 (0.009)
  Total ETDRS | 0.01 (0.054) | -0.01 (0.046)

ADVERSE EVENTS:
Time Frame: 28 Weeks
Arm/Group | High-Risk Drusen (HRD) | NCGA (Noncentral GA)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/19
Other Adverse Events (participants affected / at risk) | 21/21 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk Drusen (HRD) (N=21) | NCGA (Noncentral GA) (N=19)
Calculus urinary (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk Drusen (HRD) (N=21) | NCGA (Noncentral GA) (N=19)
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Punctate keratitis (Eye disorders) | 3 | 0
Retinal haemorrhage (Eye disorders) | 2 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Injection site pruritis (General disorders) | 21 | 17
Injection site bruising (General disorders) | 16 | 13
Injection site erythema (General disorders) | 16 | 14
Injection site induration (General disorders) | 16 | 14
Injection site pain (General disorders) | 9 | 6
Injection site haemorrhage (General disorders) | 6 | 7
Injection site urticaria (General disorders) | 5 | 4
Injection site swelling (General disorders) | 1 | 1
Injection site extravasation (General disorders) | 0 | 2
Injury associated with device (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Seasonal allergy (Immune system disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2
Procedural nausea (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Intraocular pressure increased (Investigations) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin cryotherapy (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Labile hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02848313/Prot_SAP_000.pdf